CLINICAL TRIAL: NCT07031115
Title: Linperlisib in Acquired Pure Red Cell Aplasia: a Single-arm,Cphase II Prospective Clinical Study
Brief Title: Linperlisib in the Treatment of aPRCA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Linperlisib-PRCA
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Acquired Pure Red Cell Aplasia
Keywords: Linperlisib; Acquired Pure Red Cell Aplasia; Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Linperlisib in the Treatment of aPRCA (Experimental): Linperlisib 40 mg, orally, once daily. Following 2 weeks of treatment, efficacy was assessed. If the reticulocyte count remained <20×10⁹/L, the dose was escalated to 60 mg, once daily. After an additional 2 weeks of therapy, a second efficacy assessment was performed. Patients failing to achieve partial response (PR) underwent further dose escalation to 80 mg, once daily. Treatment was discontinued if PR was not attained after 8 weeks at the maximum dose. Responding patients maintained therapy at their effective dose level. The core study period comprised 12 weeks, with responders continuing treatment at the investigator's discretion.
  Interventions: Drug: Linperlisib

INTERVENTIONS:
Drug: Linperlisib — Linperlisib 40 mg, orally, once daily. Following 2 weeks of treatment, efficacy was assessed. If the reticulocyte count remained <20×10⁹/L, the dose was escalated to 60 mg, once daily. After an additional 2 weeks of therapy, a second efficacy assessment was performed. Patients failing to achieve partial response (PR) underwent further dose escalation to 80 mg, once daily. Treatment was discontinued if PR was not attained after 8 weeks at the maximum dose. Responding patients maintained therapy at their effective dose level. The core study period comprised 12 weeks, with responders continuing treatment at the investigator's discretion.

SUMMARY:
Pure red cell aplasia (PRCA) is a syndrome characterized by normocytic normochromic anemia, reticulocytopenia, and reduced erythroid precursors in an otherwise normocellular bone marrow. It primarily affects erythropoiesis, while granulocytic and megakaryocytic lineages typically remain unaffected. First-line therapies for PRCA include corticosteroids (CS) and cyclosporine A（CsA). Although CS demonstrates high response rates, relapse frequently occurs upon dose reduction or discontinuation. CsA achieves response rates of 65%-87%, yet exhibits a delayed onset of action, often requiring 2-3 months to achieve transfusion independence. Sirolimus constitutes a second-line option, with additional therapeutic agents including methotrexate and cyclophosphamide.

Phosphatidylinositol 3-kinases (PI3Ks) represent a family of lipid kinases. The δ and γ isoforms are predominantly expressed in leukocytes and are frequently activated in various B-cell lymphomas, serving as the primary therapeutic targets for currently approved PI3K inhibitors in hematological malignancies. PI3K also plays a critical role in modulating cells of both the adaptive and innate immune systems. Studies indicate that engagement of multiple immune receptors on leukocytes triggers PI3K activation. Consequently, isoform-selective (δ or γ) or dual δ/γ inhibitors are being investigated for autoimmune conditions such as COPD, asthma, allergies, and Sjögren's syndrome. Leniolisib, the first oral PI3Kδ inhibitor approved by the FDA for immunodeficiency, exemplifies this therapeutic strategy. Several other PI3K-targeting agents are under clinical evaluation, including Parsaclisib (Phase II trial in relapsed/refractory autoimmune hemolytic anemia) and Linperlisib (Phase I trial in relapsed/refractory AIHA).

T-lymphocyte dysfunction is a pivotal factor in PRCA pathogenesis. RNA sequencing analyses have revealed significant upregulation of genes associated with the PI3K/AKT/mTOR pathway in bone marrow CD8+ T lymphocytes of patients with acquired PRCA, suggesting that targeting this pathway may represent a novel therapeutic strategy. Linperlisib, a highly selective PI3Kδ inhibitor approved for relapsed/refractory follicular lymphoma, suppresses PI3Kδ protein expression and reduces AKT phosphorylation, thereby inducing apoptosis and inhibiting lymphocyte proliferation. In 2024, a seminal report documented rapid responses and manageable tolerability with Linperlisib in four patients with acquired PRCA.

Currently, no cohort studies have been conducted on Linperlisib for PRCA treatment. This study seeks to characterize the dosing regimen, efficacy, and safety profile of Linperlisib in relapsed/refractory pure red cell aplasia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients meeting the diagnostic criteria for acquired PRCA;
* Patients who are relapsed or refractory after at least two lines of prior therapy. Refractory is defined as failure to achieve partial remission after 3 months of treatment at a stable dose of immunosuppressive agents.
* Hb ≤ 100 g/L;
* Patients with complete clinical data, demonstrated good treatment compliance, and who have signed the informed consent form;
* If taking glucocorticoids, must have discontinued them or been on a stable low maintenance dose (prednisone ≤ 15 mg/day) for at least 2 weeks prior to enrollment, and continue this dose;
* If taking immunosuppressive agents such as cyclosporine or sirolimus, must have been on a stable dose for at least 3 months, and discontinue them upon enrollment.

Exclusion Criteria:

* Patients with organ dysfunction (e.g., heart, liver, or lung) or acute renal insufficiency;
* Patients who have used PI3Kδ inhibitors within the past 6 months;
* Patients with severe infectious diseases;
* Patients with malignant tumors;
* Patients with psychiatric disorders or cognitive impairment;
* Pregnant or lactating women;
* Patients who have participated in other clinical trials within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate(ORR) | 12weeks
  ORR defined as the proportion of patients who met the criteria of either complete response (CR) or partial responce (PR).
Complete response rate (CRR) | 12weeks
  CRR defined as the proportion of patients who met the criteria of complete response.
Partial response (PR) | 12weeks
  PR defined as the patients who met the criteria of partial responce.
No response (NR) | 12weeks
  NR defined as the patients who had transfusion dependence or failed to achieve PR.

SECONDARY OUTCOMES:
Relapse rate | 12weeks
  Relapse rate defined as the proportion of patients whose response shift from PR or CR to NR
Adverse events | 12weeks
  Safety analyses include the incidence, severity grading, and dose relationship of adverse events, along with the proportion of treatment discontinuations or dose reductions due to toxicity. All adverse events that occurred or worsened during the treatment period will be reported, including those occurred later but are considered by the investigator to be related to the trial drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Means RT Jr. Pure red cell aplasia. Blood. 2016 Nov 24;128(21):2504-2509. doi: 10.1182/blood-2016-05-717140. PMID 27881371
- [Background] Sawada K, Fujishima N, Hirokawa M. Acquired pure red cell aplasia: updated review of treatment. Br J Haematol. 2008 Aug;142(4):505-14. doi: 10.1111/j.1365-2141.2008.07216.x. Epub 2008 May 28. PMID 18510682
- [Background] Mangla A, Hamad H. Pure Red Cell Aplasia. 2024 Feb 24. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK549833/ PMID 31751023
- [Background] Clark DA, Dessypris EN, Krantz SB. Studies on pure red cell aplasia. XI. Results of immunosuppressive treatment of 37 patients. Blood. 1984 Feb;63(2):277-86. PMID 6581839
- [Background] Sawada K, Hirokawa M, Fujishima N, Teramura M, Bessho M, Dan K, Tsurumi H, Nakao S, Urabe A, Omine M, Ozawa K; PRCA Collaborative Study Group. Long-term outcome of patients with acquired primary idiopathic pure red cell aplasia receiving cyclosporine A. A nationwide cohort study in Japan for the PRCA Collaborative Study Group. Haematologica. 2007 Aug;92(8):1021-8. doi: 10.3324/haematol.11192. Epub 2007 Jul 20. PMID 17640861
- [Background] Liu Y, Liu M, He X, Yang L, Zhang M, Tang P, Xing L, Niu H, Wang H. Molecular landscape of CD8+ T cells in pure red cell aplasia. Ann Hematol. 2025 Feb;104(2):953-961. doi: 10.1007/s00277-025-06220-5. PMID 39888354
- [Background] Fruman DA, Chiu H, Hopkins BD, Bagrodia S, Cantley LC, Abraham RT. The PI3K Pathway in Human Disease. Cell. 2017 Aug 10;170(4):605-635. doi: 10.1016/j.cell.2017.07.029. PMID 28802037
- [Background] Wang Z, Jiang B, Song L, Sun M, Li C, Li X, Zheng W, Tao Y, Sun Q, Qi J. Patients with acquired pure red cell aplasia respond to PI3Kdelta inhibitor rapidly. Am J Hematol. 2024 Jul;99(7):1431-1433. doi: 10.1002/ajh.27325. Epub 2024 Apr 12. No abstract available. PMID 38607227
- [Background] Red Blood Cell Disease (Anemia) Group, Chinese Society of Hematology, Chinese Medical Association. [Chinese expert consensus on the diagnosis and treatment of acquired pure red cell aplasia (2020)]. Zhonghua Xue Ye Xue Za Zhi. 2020 Mar 14;41(3):177-184. doi: 10.3760/cma.j.issn.0253-2727.2020.03.001. No abstract available. Chinese. PMID 32311886
- [Background] Hirokawa M, Sawada K, Fujishima N, Teramura M, Bessho M, Dan K, Tsurumi H, Nakao S, Urabe A, Fujisawa S, Yonemura Y, Kawano F, Oshimi K, Sugimoto K, Matsuda A, Karasawa M, Arai A, Komatsu N, Harigae H, Omine M, Ozawa K, Kurokawa M; PRCA Collaborative Study Group. Long-term outcome of patients with acquired chronic pure red cell aplasia (PRCA) following immunosuppressive therapy: a final report of the nationwide cohort study in 2004/2006 by the Japan PRCA collaborative study group. Br J Haematol. 2015 Jun;169(6):879-86. doi: 10.1111/bjh.13376. Epub 2015 Mar 25. PMID 25807974